CLINICAL TRIAL: NCT01276093
Title: Pulmonary Vein Ablation Versus Amiodarone in the Elderly
Acronym: PAVANE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: DSMB recommendation; enrollment too slow
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AF-10-023-ND-AB
Record Dates: First submitted 2011-01-11; First posted 2011-01-13 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; PVI ablation; Elderly patients; Efficacy
MeSH Terms: conditions — Atrial Fibrillation | interventions — Amiodarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PVI ablation (Experimental): Pulmonary Vein Ablation
  Interventions: Procedure: PVI ablation
- Amiodarone medical treatment (Active Comparator): Amiodarone medical treatment
  Interventions: Drug: Amiodarone

INTERVENTIONS:
Procedure: PVI ablation — Pulmonary Vein Ablation using RF.
  Other Names: Pulmonary Vein Isolation
  Arms: PVI ablation
Drug: Amiodarone — Amiodarone tablets
  Arms: Amiodarone medical treatment

SUMMARY:
The purpose of the study is to demonstrate that in patients of 70 years or older with symptomatic paroxysmal atrial fibrillation (AF) pulmonary vein isolation (PVI) using RF ablation therapy is superior to medical treatment with amiodarone to prevent recurrence of AF.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common arrhythmia. The prevalence of AF is highly age dependent as 70% of AF patients is between 65 and 85 years old. With increasing life expectancy, AF prevalence will increase 2,5 times during the next 50 years and constitute an even more important health concern. In younger patients Pulmonary vein ablation is an accepted procedure with superior efficacy compared to medical treatment. In this study the safety and efficacy of PVI in patients over 70 years old will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years at moment of screening, able to sign informed consent.
* Documented paroxysmal AF in association with complaints in the last year, with at least 2 episodes of complaints attributed to AF in the previous 2 months.
* Paroxysmal AF documented with at least one ECG with sinus rhythm not after cardioversion in the last year.
* No prior use of amiodarone in the last 6 months and no usage longer than 4 weeks in total.

Exclusion Criteria:

* EF < 35 % or description of "poor left ventricular function" on echocardiogram. Measurement should not be older than 6 months at moment of screening.
* Aortic, mitral, pulmonary or tricuspid valve regurgitation or stenosis, if graded severe (grade >3)
* Acute illness: unstable angina, infectious disease.
* Primary structural or electrical heart disease: dilated cardiomyopathy, hypertrophic cardiomyopathy, Brugada syndrome, long QT syndrome.
* Reversible causes (thyroid dysfunction, uncontrolled hypertension, ischemia).
* Previous ablation.
* Contraindications for amiodarone; liver dysfunction (serum alanine aminotransferase >2.5 times upper limit); thyroid dysfunction; chronic lung disease; baseline QTc >460 ms. sinus node dysfunction (pause more than 3 seconds in sinus rhythm); second or third degree AV-block.
* Contraindications for anti-coagulation: prior life threatening hemorrhage under use of Vitamin K antagonists.
* Any myocardial infarction or PCI in previous 6 months.
* CABG in previous 6 months.
* Renal dysfunction: creatinine clearance <45 ml/min
* Severe co-morbidity. Life expectancy less than 1 year.
* Thrombus in left atrium
* Untreatable allergy to contrast media

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 59 (Actual)
Dates: Start 2011-07; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Recurrence of episodes of AF, atypical atrial flutter or left sided atrial tachycardia | Until 1 year after post treatment blanking period

SECONDARY OUTCOMES:
Composite end point of hospitalization, stroke, major bleeding and death | Until last patient has been followed for 15 months after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Dekker, Dr, Principal Investigator — Catharina Ziekenhuis Eindhoven
Locations (6):
- Netherlands (6):
  - Elkerliek Hospital, Helmond, North Brabant
  - Maxima Medical Center, Veldhoven, North Brabant
  - Haga Hospital, The Hague, South Holland
  - Onze Lieve Vrouwen Gasthuis, Amsterdam
  - Catharina Ziekenhuis, Eindhoven
  - Medisch Spectrum Twente, Enschede